CLINICAL TRIAL: NCT03393689
Title: Kan tumorvækst Forudsiges Ved RGD-PET/MR af Vestibularis Schwannomer?
Brief Title: RGD PET/MRI in Sporadic Vestibular Schwannoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hjalte Sass, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCT2017-1; 2017-002604-27 (EudraCT Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-08 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Acoustic Neuroma
Keywords: 68Ga-NODAGA-E[c(RGDyK)]2; Angiogenesis PET/MR; Acoustic Neuroma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Angiogenesis PET/MR (Experimental): One injection of the radioligand 68Ga-NODAGA-E[c(RGDyK)]2 followed by PET/MR
  Interventions: Drug: One injection of 68Ga-NODAGA-E[c(RGDyK)]2

INTERVENTIONS:
Drug: One injection of 68Ga-NODAGA-E[c(RGDyK)]2 — One injection of 68Ga-NODAGA-E[c(RGDyK)]2

SUMMARY:
The aim of this non-randomised, prospective study is to investigate the applicability and prognostic value of angiogenesis PET/MR with the radioligand 68Ga-NODAGA- E[c(RGDyK)]2 in patients with sporadic Vestibuarl Schwannomas.

DETAILED DESCRIPTION:
The radioligand 68Ga-NODAGA- E[c(RGDyK)]2 targets the Arg-Gly-Asp (RGD) sequence known to bind with the αvβ3 integrin that is expressed on the surface of angiogenic blood vessels or tumor cells. The radioligand can be used to visualize tumor angiogenesis using PET/MR.

A total of 40 patients diagnosed with sporadic vestibular schwannomas will be subjected to an angiogenesis-PET/MR scan. Follow-up MR-only scan will be performed (from the time of the angiogenesis PET/MR) minimum 2 months later in regards to calculate growth rate. The uptake of 68Ga-NODAGA-E[c(RGDyK)]2 (Standardized Uptake Values, SUVmax) in tumor lesions will be quantified as Standardized Uptake Values (SUVmax/SUVmean) and compared with PFS, DSS and OS (dichotomized above/below median SUVmax and analyzed by Kaplan-Meier).

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years with MRI verified sporadic vestibular schwannomas
* Patients > 18 år whom max has been in watchful waiting regime in 12 months and/or max. received 1 follow-up MRI scan.
* Must be able to read and understand the patient information in Danish and to give informed consent

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Weight more than the maximum weight limit for the PET/MR bed of the scanner (140 kg)
* History of allergic reaction attributable to compounds of similar chemical or biologic composition to 68Ga-NODAGA-E[c(RGDyK)]2
* Recent systemic treatment with steroids
* Hormone treatment incl. birth control pills.
* Claustrofobia
* Non-MRI compatible implants.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-01-02 (Estimated); Study Completion 2021-01-02 (Estimated)

PRIMARY OUTCOMES:
Angiogenesis PET/MR imaging of patients with sporadic Vestibular Schwannomas | 1 hour
  The radioligand 68Ga-NODAGA-E[c(RGDyK)]2 can be used as a prognostic marker for growth rate in patients with sporadic vestibular schwannomas.

CONTACTS AND LOCATIONS:
Overall Officials: Hjalte C.R. Sass, MD, Ph.d.-Fellow, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Otolaryngology, Head and Neck Surgery & Audiology, Rigshospitalet, Copenhagen, Denmark